CLINICAL TRIAL: NCT02704338
Title: Phase 1 Clinical Trial Using Regulatory T Cells as Individualized Medicine to Evaluate the Safety and Efficacy in Autoimmune Hepatitis
Brief Title: Safety and Efficacy Study of Regulatory T Cells in Treating Autoimmune Hepatitis
Acronym: Treg
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ling Lu, Principal Investigator, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NJLT002
Record Dates: First submitted 2016-02-28; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Autoimmune Diseases
Keywords: Autoimmune Diseases, Treg
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regulatory T cells (Experimental): CD4(cluster of differentiation)+CD25+CD127- T cells isolated from peripheral blood mononuclear cells were be expanded with GMP(Good Manufacturing Practice) anti-CD3/CD28 coated beads in the presence of IL-2 and all-trans retinoid acid.
  Interventions: Biological: Regulatory T cells

INTERVENTIONS:
Biological: Regulatory T cells — Regulatory t cells will be injected back to autoimmune hepatitis patients

SUMMARY:
Separated and expanded the CD4+CD25+CD127- Tregs from peripheral blood of autoimmune hepatitis patients and administrate the cells (5 x 106 cells/kg) into patients.

DETAILED DESCRIPTION:
The trial will be carried out in autoimmune patients. The investigators will isolate CD4(cluster of differentiation)+CD25(cluster of differentiation25)+CD127(cluster of differentiation127)- Tregs from these patients, and expand them with IL(interleukin)-2 retinoid acid and anti-CD3(cluster of differentiation 3) /CD28(cluster of differentiation 28) beads. The patients will be subsequently treated with single infusion of CD4+CD25+CD127- Tregs (10-20 x 106 cells/kg).

In the clinical trials, the investigators will monitor the number of Tregs in patients at different periods, and to test their suppressive functions in vitro. Also the function and biopsy of liver will be processed to determine the efficacy of Treg therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Autoimmune hepatitis(according to the criteria defined by the international autoimmune hepatitis Group ,Hepatology, 2008;48:169-176)
3. Negative pregnancy test
4. Moderately active disease under standard treatment

Exclusion Criteria:

1. Hepatocellular carcinoma or other Malignancies
2. Pregnant or lactating women
3. Vital organs failure (Cardiac, Renal or Respiratory, et al)
4. Sepsis
5. Active thrombosis in the portal or hepatic veins
6. Concomitant psychiatric disease or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give informed consent
7. Surgery during the last 2 months or surgery planned during the study,
8. Participation in other biomedical research in the last 3 months or planned during the study.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission(serum levels of alanine aminotransferase, aspartate aminotransferase and Total bilirubin within normal ranges) | 12 months
immunology remission(=serum levels of T cell subsets, immune globulin, and complement within normal ranges) and lack of other side effects. | 12 months

SECONDARY OUTCOMES:
Incidence of biochemical remission 2 times increase of serum levels of alanine aminotransferase, aspartate aminotransferase and Total bilirubin. | 12 months
Suspected rejection detected by clinical feature or biopsy. | 12 months
Incidence of 2 times increase of immunology related level(serum levels of T cell subsets,immune globulin) or present other side effects. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wang, M.D.,PH.D., Study Chair — Nanjing Medical University

REFERENCES:
- [Derived] Chung YY, Rahim MN, Heneghan MA. Autoimmune hepatitis and pregnancy: considerations for the clinician. Expert Rev Clin Immunol. 2022 Apr;18(4):325-333. doi: 10.1080/1744666X.2022.2044307. Epub 2022 Mar 2. PMID 35179437